CLINICAL TRIAL: NCT04428671
Title: Pilot Study of Neoadjuvant/Adjuvant Cemiplimab for High Risk Cutaneous Squamous Cell Carcinoma
Brief Title: Cemiplimab Before and After Surgery for the Treatment of High Risk Cutaneous Squamous Cell Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Lowe, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00115160; NCI-2019-07373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00115160; Winship4851-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Skin Squamous Cell Carcinoma; Recurrent Skin Squamous Cell Carcinoma
MeSH Terms: interventions — cemiplimab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cemiplimab) (Experimental): NEOADJUVANT PHASE: Prior to standard of care surgery, patients receive cemiplimab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  ADJUVANT PHASE: Within 2-6 weeks after standard of care radiation therapy (or surgery if no radiation therapy), patients receive cemiplimab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cemiplimab; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN2810
Radiation: Radiation Therapy — Undergo standard of care radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery

SUMMARY:
This phase I trial studies how well cemiplimab before and after surgery works in treating patients with high risk cutaneous squamous cell cancer. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cemiplimab before surgery may improve risk of the cancer returning in patients with high risk cutaneous squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the pathologic response rate of neoadjuvant cemiplimab in cutaneous squamous cell carcinoma (cSCC).

SECONDARY OBJECTIVES:

I. To document the local recurrence rate of high-risk cSCC treated with adjuvant cemiplimab.

II. To document the systemic recurrence rate of high-risk cSCC treated with adjuvant cemiplimab.

III. To document the 6-month, 12-month, 2-year overall survival (OS), recurrence-free survival (RFS) for patients with high risk cSCC.

TERTIARY/EXPLORATORY OBJECTIVE:

I. To evaluate the immune profile of fresh tumor tissue, blood in patients with cSCC treated with cemiplimab.

OUTLINE:

NEOADJUVANT PHASE: Prior to standard of care surgery, patients receive cemiplimab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

ADJUVANT PHASE: Within 2-6 weeks after completion of standard of care radiation therapy (or surgery if no radiation therapy), patients receive cemiplimab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 2 years, every 6 months for the next 3 years, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a known diagnosis of high risk cSCC defined by the following criteria:

  * Nodal disease with extracapsular extension (ECE) and at least one node >= 20 mm on the surgical pathology report
  * In-transit metastases (ITM) defined as skin or subcutaneous metastases that are > 2 cm from the primary lesion but are not beyond the regional nodal basin
  * T4 lesion for head and neck CSCC
  * Perineural invasion (PNI), defined as clinical and/or radiologic involvement of named nerves
  * Recurrent CSCC, defined as CSCC that arises within the area of the previously resected tumor, or at least one of the following additional features:

    * >= N2b disease associated with the recurrent lesion
    * Nominal >= T3 (recurrent lesion >= 4 cm in diameter or minor bone erosion or deep invasion > 6 mm measured from the granular layer of normal adjacent epithelium)
    * Poorly differentiated histology and >= 20 mm diameter of recurrent lesion. The recurrent lesion must be documented to be within the area of the previously resected CSCC by radial measurement of the greatest radius of the final defect, measured from the estimated center of the original surgical wound
* Cancer confirmed to be surgically resectable, with surgery evaluation with planned prior to resection
* No prior systemic immunotherapy, no prior anti-PD1 therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Hemoglobin >= 9.0 g/dl (within 28 days of cycle 1 day 1)
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 28 days of cycle 1 day 1)
* Platelets >= 100,000/mcL (within 28 days of cycle 1 day 1)
* Total bilirubin =<1.5 institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 institutional upper limit of normal (ULN) (within 28 days of cycle 1 day 1)
* Albumin >= 3.0 g/dL (within 28 days of cycle 1 day 1)
* Serum creatinine =< 1.5 x ULN (or calculated creatinine clearance of >= 50 mL/min using Cockcroft-Gault formula) (within 28 days of cycle 1 day 1)
* International normalized ratio (INR) =< 1.5 (within 28 days of cycle 1 day 1)

  * Anticoagulation is allowed only with low molecular weight heparin (LMWH). Patient receiving LMW heparin on stable therapeutic dose for more than 2 weeks or with factor Xa level < 1.1U/mL are allowed on the trial
* Clinically significant toxic effect(s) of the most recent prior anti-cancer therapy must be grade 1 or resolved (except alopecia and sensory neuropathy); patients with grade 2 adrenal insufficiency related to prior anti-cancer therapy (defined as requiring medical intervention, such as concomitant steroids) or grade 2 hypothyroidism (defined as requiring hormone replacement therapy) may be enrolled provided that clinical symptoms are adequately controlled and the daily dose is 10 mg or less of prednisone or equivalent. If the patient received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of cemiplimab on the developing human fetus are unknown. For this reason female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy
* FCBP and men must agree to use adequate contraception (at least one highly effective method and one additional method of birth control at the same time or complete abstinence) prior to study entry, for the duration of study participation and for at least 6 months following study drug discontinuation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. A female of childbearing potential (FCBP) is a sexually mature woman who: has not undergone a hysterectomy or bilateral oophorectomy or has not been naturally postmenopausal for at least 12 consecutive months (if age >= 55 years); if the female subject is < 55 years and she has been naturally postmenopausal for >= 1 year her reproductive status has to be verified by additional lab tests (< 20 estradiol OR estradiol < 40 with follicle stimulating hormone [FSH] > 40 in women not on estrogen replacement therapy)
* Patients must agree not to donate blood, sperm/ova while taking protocol therapy and for at least 6 months after stopping treatment
* Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation

Exclusion Criteria:

* Determined not to be a surgical candidate due to medical co-morbidities or extent of disease
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation)
* Prior organ allograft or allogeneic bone marrow transplantation
* Subjects with active or history of immune mediated pneumonitis, colitis, hepatitis, nephritis, or skin reactions as these patients may be at increased risk for developing immune therapy-induced exacerbation or recurrence of their immune mediated disease, potentially delaying surgery
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Women who are pregnant or lactating
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Clinical evidence of bleeding diathesis or coagulopathy
* Subjects with a history of severe allergic reactions
* Patients with prior malignancies, are eligible if they have been disease free for > 3 years
* Patients with prior low-risk non-melanoma skin cancers and in situ carcinomas are eligible provided there was complete removal
* Use of other investigational drugs (drugs not marked for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Non-oncology vaccines within 28 days prior to starting treatment
* Prisoners and subjects who are compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate | From screening up to 10 years post-treatment
  Defined as the number of complete and partial responses divided by the total number of patients, as assessed by pathology. Pathological complete response (pCR) (no viable tumor) or pathological partial response (pPR) (less than 50% viable tumor) as well as near pCR (less than 10% viable tumor) in the tumor bed will be documented by pathology from the resection specimen. Pathologic response rate will be summarized using frequency and percentage, and a 95% exact confidence interval will be reported using the Clopper-Pearson method.

SECONDARY OUTCOMES:
Time to local recurrence | From screening to local recurrence, death, or last known follow-up, assessed up to 10 years post-treatment
  Local recurrence-free survival will be estimated using the Kaplan-Meier method.
Time to systemic recurrence | From screening to systemic recurrence, death, or last known follow-up, assessed up to 10 years post-treatment
  Systemic recurrence-free survival will be estimated using the Kaplan-Meier method.
Overall survival (OS) | From screening to death from any cause or last known follow-up, assessed up to 2 years post-treatment
  OS will be estimated using the Kaplan-Meier method. 6-month, 12-month, and 24-month OS estimates will be reported along with 95% confidence intervals.
Recurrence-free survival (RFS) | From screening to recurrence, death, or last known follow-up, assessed up to 2 years post-treatment
  RFS will be estimated using the Kaplan-Meier method. 6-month, 12-month, and 24-month RFS estimates will be reported along with 95% confidence intervals.

OTHER OUTCOMES:
Change in immune system biomarkers | From baseline up to 10 years post-treatment
  Pre- and post-surgery assessments of biomarkers extracted from tissue and blood samples will be summarized using frequencies and percentages for categorical variables, and mean, median, standard deviation, and range for numeric variables. Pre- versus (vs.) post-surgery values will be compared using paired t-tests or McNemar's tests, where appropriate. Biomarkers extracted from blood samples will also be collected at progression or completion of adjuvant therapy. In those cases, mixed models with a random intercept will be explored to assess the impact of time on change in biomarker status. Change in biomarker will be compared across response (yes/no) using two-sample t-tests or Mann Whitney U tests, where appropriate, and the and the impact of pre-surgery, post-surgery, and change in biomarker will be compared across survival endpoints using log-rank tests and univariate Cox proportional hazards models.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lowe, MD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.